CLINICAL TRIAL: NCT06181305
Title: Hormonal Replacement Therapy Plus Letrozole Incorporation Versus Letrozole Mild Ovarian Stimulation in Endometrial Preparation for Frozen Embryo Transfer: A Randomised Controlled Trial
Brief Title: Endometrial Preparation in Frozen Embryo Transfer Cycles
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Rahem Fertility Center (Other)
Responsible Party: Principal Investigator, Eman Elgindy, doctor, Rahem Fertility Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: endometrial preparation
Record Dates: First submitted 2023-12-12; First posted 2023-12-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: IVF
MeSH Terms: interventions — Estradiol; Letrozole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (HRT plus letrozole incorporation) (Experimental): Exogenous oestradiol in the form of 2 mg oral oestradiol valerate , three times daily will be started on the 2nd or 3rd day of the cycle. Tri-laminar endometrium of ≥ 9 mm will be the targeted cut-off. If the endometrium does not yet reach the target, oestradiol supplementation will be continued with serial US assessment until the targeted cut-off will be reached. Upon reaching the target endometrium, oral letrozole tablets 2.5 mg will be started twice daily for 5 days only with continuation of 6 mg daily oestradiol supplementation. Then, daily intramuscular progesterone in oil (100 mg intramuscular progesterone) will be started once per day with continuation of 6 mg oestradiol
  interventions:
  Drug:estradiol valertae
  Drug :letrozole 2.5 mg tablet
  Interventions: Drug: estradiol valerate and letrozole
- Group B (Letrozole mild ovarian stimulation) (Active Comparator): Oral letrozole 2.5-5 mg daily on cycle day(3-7) will be added . TVS will be performed from cycle day 8-10 to make sure that a dominant follicle has been recruited with the endometrium thickness ≥ 7 mm . Upon reaching the dominant follicle (18-20mm) , endometrial thickness will be measured on the day of ovulation trigger and blood sample will be withdrawn from each patient for assessment of E2 , P4 and LH levels. Patients with low LH level , high E2 level , low P4 level (<1 ng/ml) will continue in the RCT; 10,000unit HCG will be injected as ovulation trigger
  intervention :
  Drug :letrozole 2.5mg tablet
  procedure: on the day of ovulation trigger blood sample will be withdrawn from each patient for assessment of E2 , P4 and LH levels.
  Interventions: Drug: letrozole 2,5 mg tablet

INTERVENTIONS:
Drug: estradiol valerate and letrozole — hormone replacement therapy by estradiol valerate plus letrozole incorporation .
  Arms: Group A (HRT plus letrozole incorporation)
Drug: letrozole 2,5 mg tablet — mild ovarian stimulation
  Arms: Group B (Letrozole mild ovarian stimulation)

SUMMARY:
In order to get optimal pregnancy rates after frozen embryo transfer (FET), the embryo stage and endometrium should be synchronized. Endometrial preparation is done by either natural, artificial (Hormonal replacement therapy HRT) , modified natural methods or mild ovarian stimulation. HRT cycle has a better schedualization however, there are some reports about higher rates of miscarriage, pregnancy induced hypertension (PIH) and preeclampsia (PET) in HRT cycles. A recent study has found that incorporation of the aromatase inhibitor (letrozole) to HRT cycles was associated with better FET outcomes in comparison to hormonal replacement therapy cycles alone. Meanwhile, mild ovarian stimulation protocol can be done either by oral drugs like letrozole or by letrozole plus gonadotropins . So this study aims to compare the reproductive outcomes in two endometrial preparation protocols for frozen embryo transfer cycles; letrozole mild ovarian stimulation versus HRT plus letrozole incorporation.

DETAILED DESCRIPTION:
In order to get optimal pregnancy rates after frozen embryo transfer (FET), the embryo stage and endometrium should be synchronized. This can be done by hormonal replacement therapy (HRT), natural cycles (NC), modified natural cycles or mild ovarian stimulation. In hormonal replacement therapy cycle, estrogen and progesterone are sequentially given to resemble the hormonal course of the natural cycle . Hormonal replacement therapy cycle has a better schedualization and is used for patients with irregular cycles as polycystic ovary syndrome ( PCOS). However, there are some reports about higher rates of miscarriage, pregnancy induced hypertension (PIH) and preeclampsia (PET) in HRT cycles.

A recent study has found that incorporation of the aromatase inhibitor (letrozole) to HRT cycles was associated with better FET outcomes in comparison to HRT cycles alone. Ongoing pregnancy rate (OPR) was higher in HRT plus letrozole group than HRT only group.

Letrozole is a third-generation aromatase inhibitor that leads to mono-ovulatory cycles with short half-life . Miller and his colleagues found that letrozole increased Integrin expression and improved pregnancy and implantation rates among women with endometrial receptivity defects . Another study found that ovarian stimulation with letrozole was associated with increase in the expression of uterine receptivity markers including integrin, leukemia inhibitory factor, and L-selectin.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 18 and 37 years with either regular cycles or oligomenorrhoea or amenorrhoea.
* Women undergoing FET cycles.
* Participants should have at least one good-quality blastocyst available for vitrification and also for transfer after warming.
* Participants having optimal endometrium before starting luteal phase support

Exclusion Criteria:

* Women who will refuse to participate in in the study.
* Women who will not reach the optimal endometrium.
* Participants that don't have at least one good-quality blastocyst for transfer after warming.
* PGT embryos will be excluded.

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 210 (Estimated)
Dates: Start 2024-02-24 (Actual); Primary Completion 2024-11-25 (Estimated); Study Completion 2024-12-25 (Estimated)

PRIMARY OUTCOMES:
ongoing pregnancy rate (OPR) | 12 weeks
  Number of pregnant women with viable fetus at 12 weeks gestation per woman randomized

SECONDARY OUTCOMES:
Clinical pregnancy rate (CPR) | 5 weeks after embryo transfer
  Number of gestational sacs with evident fetal pulsations per woman randomized,ectopic pregnancy is also includded pregnancy is aslo included
Ectopic pregnancy | 7 week
  pregnancy outside the uterine cavity diagnosed by ultrasound ,surgical visualization or histopathology
Miscarriage rate | 12 weeks
  Number of miscarriages per woman with positive pregnancy tests
Implantation rate | 21 days after embryo transfer
  Number of gestational sac recognized by ultrasound in uterus 3 weeks after embryo transfer
live birth rate | 22 completed weeks of gestational age
  The complete expulsion or extraction from a woman of a product of fertilization,after 22 complete weeks of gestational age;which,after such separation,breathes or shows any other evidence of life,such as heart beat,umblical cord pulsation or definite movement of voluntary muscles,irrespective of whether the umblical cord has been cut or the placenta is attached.A birth weight of 500 grams or more can be used if gestational age is unknown.Live births refer to the individual newborn ;for example,a twin delivery represents two live births
Number of participants with Hypertensive disorders of pregnancy | 20 weeks gestation till postpartum
  gestational hypertension or preeclampsia
Number of participants with Large for gestational age | from gestation till delivery
  A birth weight greater than the 90th centile of the sex-specific birth weight for a given gestational age reference

CONTACTS AND LOCATIONS:
Overall Officials: Eman El-gindy, MD,PhD, Principal Investigator — Rahem Fertility Center
Locations (1):
- Rahem fertility center, Zagazig, Egypt

REFERENCES:
- [Background] Elgindy EA, Abdelghany AA, Sibai AbdAlsalam H, Mostafa MI. The novel incorporation of aromatase inhibitor in hormonal replacement therapy cycles: a randomized controlled trial. Reprod Biomed Online. 2022 Apr;44(4):641-649. doi: 10.1016/j.rbmo.2021.10.025. Epub 2021 Dec 20. PMID 35288021
- [Background] Ezoe K, Fukuda J, Takeshima K, Shinohara K, Kato K. Letrozole-induced endometrial preparation improved the pregnancy outcomes after frozen blastocyst transfer compared to the natural cycle: a retrospective cohort study. BMC Pregnancy Childbirth. 2022 Nov 7;22(1):824. doi: 10.1186/s12884-022-05174-0. PMID 36344952
- [Background] An BGL, Chapman M, Tilia L, Venetis C. Is there an optimal window of time for transferring single frozen-thawed euploid blastocysts? A cohort study of 1170 embryo transfers. Hum Reprod. 2022 Nov 24;37(12):2797-2807. doi: 10.1093/humrep/deac227. PMID 36305795
- [Background] Mumusoglu S, Polat M, Ozbek IY, Bozdag G, Papanikolaou EG, Esteves SC, Humaidan P, Yarali H. Preparation of the Endometrium for Frozen Embryo Transfer: A Systematic Review. Front Endocrinol (Lausanne). 2021 Jul 9;12:688237. doi: 10.3389/fendo.2021.688237. eCollection 2021. PMID 34305815
- [Background] Zhang J, Liu H, Wang Y, Mao X, Chen Q, Fan Y, Xiao Y, Kuang Y. Letrozole use during frozen embryo transfer cycles in women with polycystic ovary syndrome. Fertil Steril. 2019 Aug;112(2):371-377. doi: 10.1016/j.fertnstert.2019.04.014. Epub 2019 May 21. PMID 31126712
- [Background] Godiwala P, Makhijani R, Bartolucci A, Grow D, Nulsen J, Benadiva C, Grady J, Engmann L. Pregnancy outcomes after frozen-thawed embryo transfer using letrozole ovulation induction, natural, or programmed cycles. Fertil Steril. 2022 Oct;118(4):690-698. doi: 10.1016/j.fertnstert.2022.06.013. Epub 2022 Jul 19. PMID 35863997
- [Background] Lawrenz B, Melado L, Fatemi HM. Frozen embryo transfers in a natural cycle: how to do it right. Curr Opin Obstet Gynecol. 2023 Jun 1;35(3):224-229. doi: 10.1097/GCO.0000000000000862. Epub 2023 Mar 14. PMID 36924405